CLINICAL TRIAL: NCT02762266
Title: International Randomized Study of Transarterial Chemoembolization (TACE) Versus Stereotactic Body Radiotherapy (SBRT) / Stereotactic Ablative Radiotherapy (SABR) for Residual or Recurrent Hepatocellular Carcinoma After Initial TACE
Brief Title: Transarterial Chemoembolization Compared With Stereotactic Body Radiation Therapy or Stereotactic Ablative Radiation Therapy in Treating Patients With Residual or Recurrent Liver Cancer Undergone Initial Transarterial Chemoembolization
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision - funding
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erqi Liu Pollom, Associate Professor of Radiation Oncology (Radiation Therapy), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-35937; NCI-2016-00418 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA124435 (NIH); HEP0052 (Other: OnCore ID)
Record Dates: First submitted 2016-04-05; First posted 2016-05-04 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Child-Pugh Class A; Child-Pugh Class B; Recurrent Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; ethylene-vinyl alcohol copolymer; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (TACE) (Active Comparator): Patients undergo TACE.
  Interventions: Procedure: Transarterial Chemoembolization; Drug: embolic agent; Drug: lipiodol
- Arm II (SBRT) (Experimental): Beginning within 2 weeks of the radiation set-up scan and within 4 weeks of fiducial seed implantation (if applicable), patients undergo image guided SBRT 3 fractions within 1 week or 5 fractions within 2 weeks.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT
  Arms: Arm II (SBRT)
Procedure: Transarterial Chemoembolization — Undergo TACE
  Other Names: TACE
  Arms: Arm I (TACE)
Drug: embolic agent — . Acceptable embolic agents include:
  * Gelatin sponge (gelfoam)
  * Polyvinyl alcohol (PVA) particles
  * Microspheres / Embolic beads
  Arms: Arm I (TACE)
Drug: lipiodol
  Arms: Arm I (TACE)

SUMMARY:
This randomized phase III trial studies how well transarterial chemoembolization (TACE) works compared to stereotactic body radiation therapy (SBRT) or stereotactic ablative radiation therapy (SABR) in patients with liver cancer that remain after attempts to remove the cancer have been made (residual) or has come back (recurrent). TACE is a minimally invasive, image-guided treatment procedure that uses a catheter to deliver both chemotherapy medication and embolization materials into the blood vessels that lead to the tumors. SBRT or SABR may be able to send radiation directly to the tumor and cause less damage to normal liver tissue. It is not yet known whether TACE is more effective than SBRT or SABR in treating patients with persistent or recurrent liver cancer who have undergone initial TACE.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the freedom from local progression (FFLP) of TACE versus (vs) SABR in patients with persistent hepatocellular carcinoma (HCC) after TACE.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) of TACE vs SABR in patients with persistent HCC after initial TACE.

II. To determine the overall survival (OS) of TACE vs SABR for persistent HCC. III. To determine the toxicities associated with TACE or SABR for persistent HCC.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients undergo TACE.

ARM II: Beginning within 2 weeks of the radiation set-up scan and within 4 weeks of fiducial seed implantation (if applicable), patients undergo image guided SBRT 3 fractions within 1 week or 5 fractions within 2 weeks.

After completion of study treatment, patients are followed up for 1-2 weeks, 1, 3, 6, 12, and 18 months, and every 6 months up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hepatocellular carcinoma (HCC) by one of the following:

  * Histopathology
  * One radiographic technique that confirms a lesion >= 1 cm with arterial hypervascularization with washout on delayed phase
* Radiographic evidence of persistent, progressive, or recurrent disease in an area previously treated with TACE and determined from 3 months after initial TACE; this evaluation should be within 6 weeks of date of study eligibility
* Unifocal liver tumors not to exceed 7.5 cm in greatest axial dimension; multifocal lesions will be restricted to lesions that can be treated within a single target volume within the same liver segment and to an aggregate of 10 cm as long as the dose constraints to normal tissue can be met
* Eastern Clinical Oncology Group (ECOG) performance status 0, 1 or 2
* Patients with liver disease classified as Child Pugh class A or B, with score =< 9 ((within 4 weeks of treatment)
* Life expectancy >= 6 months
* Ability of the research subject or authorized legal representative to understand and have the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior radiotherapy to the upper abdomen
* Prior radioembolization to the liver
* Prior radiofrequency ablation (RFA) to index lesion
* Liver transplant
* Active gastrointestinal bleed within 2 weeks of study enrollment
* Ascites refractory to medical therapy (mild to moderate ascites is allowed)
* Women who are pregnant or breastfeeding
* Administration of chemotherapy within the last 1 month
* Extrahepatic metastases
* Participation in another concurrent treatment protocol
* Prior history of malignancy other than HCC, dermatologic basal cell or squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erqi Liu Pollom, MD, Principal Investigator — Stanford University; Daniel Chang, MD, Principal Investigator — Stanford University
Locations (2):
- Stanford University, School of Medicine, Palo Alto, California, United States
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 participants signed informed consent, 12 were randomized to a study arm.
Groups:
- Transarterial Chemoembolization (TACE): Patients undergo TACE using an embolic agent (gelatin sponge [gelfoam], polyvinyl alcohol particles, or embolic beads).
- Stereotactic Body Radiation Therapy (SBRT): Patients undergo image-guided SBRT (3 fractions within 1 week or 5 fractions within 2 weeks).
Period: Overall Study
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Started | 6 | 6
Received Treatment | 4 | 6
Completed | 4 | 6
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received treatment
Groups:
- Transarterial Chemoembolization (TACE): Patients undergo TACE using an embolic agent.
- Stereotactic Body Radiation Therapy (SBRT): Patients undergo image-guided SBRT.
- Total: Total of all reporting groups
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT) | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (6.25) | 67.7 (7.15) | 68.6 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 9
  Japan | 1 | 0 | 1
Elevated Serum Alpha-Fetoprotein (AFP) [Count of Participants; unit: Participants] — Population: Participants with AFP data
  Participants
    number analyzed (Participants) | 3 | 6 | 9
    (all) | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Local Progression Event
Description: Local progression event: occurring in the treated hepatic lesion.
Time Frame: Up to 12 months
Population: Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
Participants | 0 | 0

2. Secondary Outcome: Comparison of Median Freedom From Extra Hepatic Progression
Description: The time to freedom from extra hepatic progression will be estimated by competing risk models with death as a competing risk. Risk factors such as tumor size and institution will be tested in a multivariate Cox regression model adjusting for the competing risks.
Time Frame: Up to 16 weeks
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

3. Secondary Outcome: Median Extra Hepatic PFS for Patients With Tumors Smaller Than 3 cm and Greater Than 3 cm Per Treatment Group
Description: Extra hepatic PFS within each subgroup will be summarized by cumulative incidence function estimators adjusted for the competing risk of death or regional or distant progression.
Time Frame: At 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

4. Secondary Outcome: Median FFLP for Patients With Tumors Smaller Than 3 cm and With Tumors Greater Than 3 cm Per Treatment Group
Description: FFLP within each subgroup will be summarized by cumulative incidence function estimators adjusted for the competing risk of death or regional or distant progression.
Time Frame: At 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

5. Secondary Outcome: Median OS
Description: Overall survival will be summarized using Kaplan-Meier curves and medians with 95% confidence intervals calculated using Greenwood's formula. Log rank tests will be used to compare treatment groups. Cox proportional hazard models will be used to estimate hazard ratios between treatment groups and to assess other risk factors, in particular the effect of tumor size and the impact of the different institutions.
Time Frame: Time from randomization until death from any cause, assessed up to 3 years
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

6. Secondary Outcome: Median OS for Patients With Tumors Smaller Than 3 cm and Greater Than 3 cm Per Treatment Group
Description: Within each subgroup OS will be summarized using Kaplan-Meier curves and medians with 95% confidence intervals calculated using Greenwood's formula.
Time Frame: At 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

7. Secondary Outcome: Number of Participants With Disease Progression or Death
Description: Including local, regional, or distant progression events, or death. Local progression event: occurring in the treated tumor. Regional progression event: occurring in the same part of the body as the treated tumor. Distant progression event: occurring outside the region of the body where the treated tumor is located.
Time Frame: Randomization through 3 years
Population: Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
Participants | 1 | 3

8. Secondary Outcome: Number of Participants With Disease Progression or Death by Tumor Size (<= 3 cm and > 3 cm) Per Treatment Group
Description: as for outcome 7
Time Frame: Randomization through 18 months
Population: Participants who receive treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
Participants
  <= 3 cm: number analyzed (Participants) | 4 | 4
  <= 3 cm | 1 | 2
  > 3 cm: number analyzed (Participants) | 0 | 2
  > 3 cm |  | 1

9. Secondary Outcome: The Impact of Elevated Serum Alpha-Fetoprotein Level (AFP) on Freedom From Local Progression (FFLP)
Description: The impact of elevated AFP level on time to event endpoints will be evaluated both in terms of the initial AFP level and on-study levels in a Cox proportional hazards model.
Time Frame: Up to 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

10. Secondary Outcome: The Impact of Elevated Serum Alpha-Fetoprotein Level (AFP) on Progression-free Survival (PFS)
Description: as for outcome 9
Time Frame: Up to 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

11. Secondary Outcome: The Impact of Elevated Serum Alpha-Fetoprotein Level (AFP) on Extra Hepatic PFS
Description: The impact of elevated AFP level on time to event endpoints: FFLP, PFS, extra hepatic PFS and OS will be evaluated both in terms of the initial AFP level and on-study levels in a Cox proportional hazards model.
Time Frame: Up to 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

12. Secondary Outcome: The Impact of Elevated Serum Alpha-Fetoprotein Level (AFP) on Overall Survival (OS)
Description: as for outcome 9
Time Frame: Up to 18 months
Population: Participants who received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 4 | 6
months | NA [NA to NA] — Not calculable due to an insufficient number of events | NA [NA to NA] — Not calculable due to an insufficient number of events

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Transarterial Chemoembolization (TACE) | Stereotactic Body Radiation Therapy (SBRT)
All-Cause Mortality (participants affected / at risk) | 0/6 | 3/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transarterial Chemoembolization (TACE) (N=6) | Stereotactic Body Radiation Therapy (SBRT) (N=6)
Cholecystitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transarterial Chemoembolization (TACE) (N=6) | Stereotactic Body Radiation Therapy (SBRT) (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 4
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 2
Bloating (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
GI disorder other (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 3 | 3
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic Pain (Hepatobiliary disorders) | 1 | 0
Portal Hypertension (Hepatobiliary disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2
Alkaline Phosphatase increased (Investigations) | 0 | 2
ALT (Investigations) | 1 | 1
AST increased (Investigations) | 2 | 4
Blood Bilirubin increased (Investigations) | 1 | 4
Creatinine increased (Investigations) | 0 | 1
INR increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 1 | 6
WBC decreased (Investigations) | 0 | 2
(Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study did not enroll the planned number of participants and did not meet the protocol-prespecified threshold for statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT02762266/Prot_SAP_000.pdf